CLINICAL TRIAL: NCT03056092
Title: Cytokine and Visual Outcome Variations in Eyes Receiving a Variable Dosing Ranibizumab Treatment: The COVERT Study
Brief Title: Cytokine and Visual Outcome Variations in Eyes Receiving Ranibizumab
Acronym: COVERT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COVERT
Record Dates: First submitted 2017-02-01; First posted 2017-02-17 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Age Related Macular Degeneration; Diabetic Macular Edema; Macular Edema; Retinal Vein Occlusion
Keywords: ranibizumab; aqueous cytokine; age related macular degeneration; diabetic macular edema; retinal vein occlusion
MeSH Terms: conditions — Macular Degeneration; Macular Edema; Retinal Vein Occlusion

STUDY DESIGN:
Intervention Model Description: This study will include patients with 3 different diseases who will receive the same treatment (ranibizumab injections) but that will be independently analyzed. One population will be composed of patients with neovascular age related macular degeneration, the other of diabetic macular edema and the third of patients with macular edema secondary to retinal vein occlusion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- AMD/RVO/DME (Other): Patients presenting to St. Michael's Hospital retina clinic with neovascular age related macular degeneration, macular edema secondary to RVO and diabetic macular edema treated with intravitreal ranibizumab in a variable dosing regimen.
  Interventions: Drug: Intravitreal ranibizumab

INTERVENTIONS:
Drug: Intravitreal ranibizumab — Patients will be treated with intravitreal ranibizumab and have their aqueous humor obtained for cytokine analysis at every visit that an intravitreal injection is done

SUMMARY:
Objective: To determine the association between baseline aqueous cytokine levels and treatment intervals for patients under a variable dosing regimen with intravitreal ranibizumab in patients with neovascular age-related macular degeneration (nAMD), macular edema secondary to retinal vein occlusion (RVO) and diabetic macular edema (DME).

Methods: A prospective, single-centre study will be performed containing 3 sub-studies according to each study population: nAMD, macular edema secondary to RVO and DME. Inclusion criteria are: patients followed at St. Michael's Hospital with the diagnosis of nAMD, macular edema secondary to RVO or DME. Patients will be excluded if visual acuity is worse than counting fingers, with macular pathologies causing any structural changes to the retina, have received anti-VEGF injections or photocoagulation therapy 6 months prior to study, intraocular surgery 3 months prior to study, any history of vitreoretinal surgery or ocular inflammation in the study eye, use of systemic or topical anti-inflammatory or steroids, patients on dialysis for renal failure, allergy to the study drug or fluorescein, <18 years old, women who are pregnant. All patients will be treated with ranibizumab intravitreal injections on a variable dosing regimen: Patients with DME will be examined monthly and receive mandatory injection for the first three months (baseline, weeks 4 and 8). Afterwards, they will continue to be seen monthly and the need for new injections will be decided upon the clinical findings at each visit. An anterior chamber (AC) tap will be done if an injection is required at the visit. Patients with nAMD and RVO will be examined monthly and receive mandatory injection for the first three months. From weeks 12 until 72 (month 18), the visits will be scheduled at increasing 2-weeks intervals based on the stability of the ocular condition and response to treatment. At each visit, an injection and AC tap will be performed. The maximum interval in between injections is 12 weeks. If the disease becomes unstable, the interval in between injections is shortened and, once it stabilizes, the treatment frequency is extended again. In all patients, baseline aqueous humour specimens will be obtained prior to the first ranibizumab intravitreal injection and follow-up samples will be taken immediately prior to subsequent injections based on the treatment regimens for cytokine analysis in the end of the follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of active choroidal neovascularization secondary to AMD in the study eye
* Diagnosis of macular edema secondary to RVO: central macular thickness >310μm due to intraretinal or subretinal edema in the study eye as measured on OCT
* Diagnosis of DME with central macular thickness >310μm in the study eye as measured on OCT in patients with diabetes mellitus types 1 or 2

Exclusion Criteria:

* Previous intravitreal drug injections in either eye within 6 months prior to study enrollment
* Visual acuity worse than counting fingers
* Patients with other macular pathologies causing structural changes to the retina
* Patients with large submacular hemorrhages or extensive fibrosis occupying the majority (>50%) of the lesion
* Intraocular surgery in the study eye 3 months prior to study enrollment
* Previous vitreoretinal surgery in the study eye
* Previous photodynamic or macular photocoagulation therapy within the past 6 months in the study eye for patients with AMD
* Previous photocoagulation therapy within 6 months in the study eye or anticipated need for during the course of the study for patients with RVO
* Presence of active proliferative diabetic retinopathy or patients who have had pan-retinal photocoagulation within 6 months or patients where the need to pan-retinal photocoagulation is anticipated during the course of the study for patients with DME
* History of intraocular inflammation in the study eye
* Patients on systemic or topical anti-inflammatory or steroids medications
* Patients receiving dialysis for renal failure
* Known allergy to the study drug or fluorescein
* Patients who are pregnant
* Unwilling or unable to follow or comply with all study related procedures or to sign consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2017-02-28 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Association between aqueous cytokine levels and optimal treatment interval | 18 months
  Optimal treatment intervals based on aqueous cytokine levels

SECONDARY OUTCOMES:
Individualized relationships between aqueous cytokines and treatment response | 18 months
  Aqueous cytokine curves for each patient over based on the relationship between cytokine levels and treatment response
Relationship between cytokine threshold level and visual/anatomic outcomes | 18 months
  Cytokine threshold level below which visual and anatomic outcomes are greatest
Snellen visual acuity change | months 1, 2 and at every visit scheduled for each injection throughout 18 months period
  Snellen Best Corrected Visual Acuity (BCVA) change at months 1 and 2, and at the visits scheduled for each injection throughout an 18 months period
ETDRS visual acuity change | month 2, visits closest to injection of months 6, 12 and 18
  Visual acuity (ETDRS) change at month 2 (at the third injection), at the visits closest to injection of months 6, 12 and 18.
Optical coherence tomography (OCT) change | months 1 and 2, and at the visits scheduled for each injection throughout an 18 months period.
  Anatomic OCT change (Macular Volume, Central Macular Thickness) at months 1 and 2, and at the visits scheduled for each injection throughout an 18 months period.
Average number of injections needed | 18 months
  Average number of injections needed in a variable dosing regimen protocol over an 18 months period.

CONTACTS AND LOCATIONS:
Overall Officials: Rajeev Muni, Principal Investigator — Unity Health Toronto
Locations (2):
- Canada (2):
  - Department of Ophthalmology, St Michael's Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto

IPD SHARING:
Plan to Share IPD: No